CLINICAL TRIAL: NCT00390143
Title: Assess Long Term Persistence of a Primary Dose of GSK Biologicals' Meningococcal Vaccine 134612 Versus One Dose of Mencevax™ ACWY in Healthy Adolescents/Young Adults (15 to 19 Years at Vaccination)
Brief Title: Study in Adolescents/Adults to Evaluate the Persistence up to 3.5 Yrs of GSK Biologicals Meningococcal Vaccine 134612
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108595 Mth18; 108596 (Other: GSK); 108598 (Other: GSK)
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Meningococcal
Keywords: Immunogenicity; Meningococcal vaccine; Conjugate vaccine; Persistence
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Group A (Experimental): Subjects previously primed with meningococcal vaccine 134612.
  Interventions: Biological: Meningococcal vaccine 134612
- Group B (Active Comparator): Subjects previously primed with Mencevax™ ACWY.
  Interventions: Biological: Mencevax™ ACWY

INTERVENTIONS:
Biological: Meningococcal vaccine 134612 — One intramuscular dose during the primary study
  Arms: Group A
Biological: Mencevax™ ACWY — One subcutaneous dose during the primary study
  Arms: Group B

SUMMARY:
This study will investigate the long-term protection offered by GSK Biologicals' meningococcal vaccine 134612 up to 3.5 years after vaccination. Subjects were vaccinated at 15 to 19 years of age. This extension phase starts 18 months after vaccination and part of the subjects who were vaccinated in the primary study will be enrolled in this extension phase. No new subjects will be enrolled. This protocol posting deals with objectives & outcome measures of the extension phase 18, 30 and 42 months after vaccination. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT00126945). The Protocol Posting has been updated in order to comply with the FDA Amendment Act, September 2007.

DETAILED DESCRIPTION:
Subjects were previously vaccinated at 15 to 19 years of age with GSK Biologicals' meningococcal vaccine 134612 or with Mencevax™ ACWY. This extension phase starts 18 months after vaccination and part of the subjects will be enrolled in this extension phase. No additional vaccines will be administered during this study and no new subjects will be enrolled. The subjects will have three blood samples taken: at 18, 30 and 42 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol.
* A male or female, who was primed with meningococcal vaccine 134612 or Mencevax™ ACWY in the primary vaccination study 18 months before the first persistence assessment and who completed that study.
* Written informed consent obtained from the subject/ from the parent or guardians of the subject.
* Written informed assent obtained from the subject, as applicable, at the time of study entry.

Exclusion Criteria:

• Administration of a meningococcal polysaccharide or a meningococcal polysaccharide conjugate vaccine since the last visit of the primary vaccination study.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Meningococcal rSBA titres. | At the start of this persistence study and 12 and 24 months later.
Anti-meningococcal polysaccharide concentrations | At the start of this persistence study and 12 and 24 months later.
Occurrence of serious adverse events related to vaccination, adverse events related to lack of vaccine efficacy or study participation. | From the last study contact of the primary vaccination study to the end of this persistence study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ostergaard L, Van der Wielen M, Bianco V, Miller JM. Persistence of antibodies for 42 months following vaccination of adolescents with a meningococcal serogroups A, C, W-135, and Y tetanus toxoid conjugate vaccine (MenACWY-TT). Int J Infect Dis. 2013 Mar;17(3):e173-6. doi: 10.1016/j.ijid.2012.10.001. Epub 2012 Dec 13. PMID 23246368
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 108595 Mth18 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108595 Mth18 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108595 Mth18 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108595 Mth18 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108595 Mth18 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108595 Mth18 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register